CLINICAL TRIAL: NCT02863068
Title: A Phase II Study of Topical Sodium Nitrite in Patients With Sickle Cell and Leg Ulcers
Brief Title: Topical Sodium Nitrite in Sickle Cell Disease and Leg Ulcers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated prior to achieving target enrollment due to slow recruitment and high cost of obtaining new study drug. Since no additional funds were to be available due to end of the funding period, remaining funds were expended on analyses.
Sponsor: caterina P minniti (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor-Investigator, caterina P minniti, Professor, Montefiore Medical Center
Organization: Montefiore Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-6015
Record Dates: First submitted 2016-05-16; First posted 2016-08-11 (Estimated); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; sodium nitrite; wound healing; Ulcer
MeSH Terms: conditions — Anemia, Sickle Cell; Ulcer | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): patients will receive placebo and standard of care
  Interventions: Other: Placebo
- topical sodium nitrite (Experimental): patients will receive 2% topical sodium nitrite cream and standard of care
  Interventions: Drug: Topical Sodium Nitrite

INTERVENTIONS:
Drug: Topical Sodium Nitrite — Subjects will have 0.1 cm of 2% sodium nitrite cream applied per 1 cm2 of the total ulcerated area. Areas will be rounded to the nearest 1 cm2. If a subject has more than one ulcer, all of them will be treated with either "study cream" in this intervention.
  Arms: topical sodium nitrite
Other: Placebo — Subjects will have Placebo applied to total ulcerated area. If a subject has more than one ulcer, all of them will be treated with placebo in this intervention.
  Arms: control

SUMMARY:
The investigators are conducting a Phase II prospective and placebo controlled study of a topical cream containing sodium nitrite compared to the current standard of care. Sodium nitrite is a local donor of nitric oxide, which is known to improve blood flow and decrease bacterial load in the ulcer bed. The primary objectives are to evaluate the safety of topical sodium nitrite cream treatment in patients with sickle cell disease and chronic leg ulcers and to determine its effectiveness in accelerating the healing process and decreasing the pain associated with ulceration.

Potential benefit will be a durable resolution or improvement of the leg ulcer and its associated pain. Possible side effects include decreased blood pressure and methemoglobinemia, secondary to sodium nitrite absorption through the ulcerated skin.

Funding source FDA OOPD.

DETAILED DESCRIPTION:
Chronic leg ulcers are a complication of many blood disorders such as sickle cell disease, thalassemia, and other red blood cell disorders. In these disorders, red blood cells break down earlier than normal, which researchers suspect may cause or contribute to the development of leg ulcers; however, the exact cause is unknown, and current therapies are not very effective. Researchers are interested in determining if a research cream made with sodium nitrite, a substance that is known to increase blood flow by dilating blood vessels, may speed up the healing of skin ulcers.

Investigators are planning to enroll fifty patients with sickle cell disease to be randomized and treated twice a week with sodium nitrite cream or a placebo for ten weeks. The following events will be compared in treatment and placebo arms: a) changes in blood pressure; b) changes in pulse oximetry; c) changes in methemoglobin levels; d) any adverse events; e) rate of sickle cell disease (SCD) related complications; f) changes in biomarkers of inflammation and other laboratory data such as complete blood count and chemistries.

In order to determine if topical sodium nitrite accelerates wound healing and decreases pain at the wound site compared to placebo in patients receiving similar levels of wound care, investigators will a) accurately measure and photograph ulcers at baseline, after a two week run-in period and at predefined time points during the study and compare treatment arm to placebo; b) pain scores at wound sites will be recorded and compared for the two groups, c) Investigators will calculate opioid intake in the two arms and d) quality of life measures before and at the end of the trial

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of sickle cell disease (SS, SC, Sß-thalassemia, SD, SOArab)
* Have one or more ulcers of the one or both leg or foot
* Total surface area of leg ulcer(s) that will receive treatment must be no larger than 100 cm2
* No history of congenital methemoglobinemia
* Have documented normal Glucose-6-Phosphate Dehydrogenase (G6PD) activity

Exclusion Criteria:

* Exposure to therapeutic nitric oxide, L-arginine, nitroprusside or nitroglycerine within the past 1 week
* Subjects presenting with clinically diagnosed bacterial infection (e.g., osteomyelitis, pneumonia, sepsis or meningitis)
* Subjects who have a pre-existing methemoglobinemia (more than 3.5% on two different occasions)
* Patients who are currently enrolled in any other investigational drug study (this does not include observational or natural history protocols)
* Use of Phosphodiesterase type 5 (PDE5) inhibitors, such as sildenafil, 4 days prior to screening
* Pregnant women - urine or serum Human chorionic gonadotropin (hCG)+ or nursing mothers
* The following list of drugs and agents may cause methemoglobinemia and should be avoided while on this study:

Anesthetics (local): Benzocaine, procaine, prilocaine, Anbesol, Orajel Antimalarials: chloroquine, primaquine, quinacrine Aniline dyes Chlorates Dapsone Diarylsulfonylureas Doxorubicin Metoclopramide Nitric and nitrous oxide Nitrobenzenes (shoe and floor polish and in paint solvents) Nitroethane (artificial nail remover, propellant, fuel additive) Nitrofurantoin (furadantin) Pyridium (phenazopyridine) Phenacetin Phenylhydrazine Rasburicase Sulfonamides (sulfacetamide, sulfamethoxazole, sulfanilamide, sulfapyridine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Minniti, M.D., Principal Investigator — Montefiore Medical Center
Locations (3):
- United States (3):
  - Montefiore Medical Center - Albert Einstein College of Medicine, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minniti CP, Gorbach AM, Xu D, Hon YY, Delaney KM, Seidel M, Malik N, Peters-Lawrence M, Cantilena C, Nichols JS, Mendelsohn L, Conrey A, Grimes G, Kato GJ. Topical sodium nitrite for chronic leg ulcers in patients with sickle cell anaemia: a phase 1 dose-finding safety and tolerability trial. Lancet Haematol. 2014 Dec 1;1(3):e95-e103. doi: 10.1016/s2352-3026(14)00019-2. PMID 25938131

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 patients (pts) were screened and 24 consented (one was consented twice as the IRB required a reconsent due to the time interval which had lapsed between the consent process and study initiation during COVID). Of the 24 unique pts, 2 were lost to follow up during the run-in period and 4 pts had a reduction in ulcer size by >25%, via normal wound care, during the run-in period and were not eligible for study-defined treatment and not enrolled into the study. As such, 18 pts were enrolled.
Groups:
- Placebo: Participants will receive placebo and standard of care
  Placebo: Participants will have Placebo applied to total ulcerated area. If a participant has more than one ulcer, all of them will be treated with placebo in this intervention.
- Topical Sodium Nitrite: Participants will receive 2% topical sodium nitrite cream and standard of care
  Topical Sodium Nitrite: Participants will have 0.1 cm of 2% sodium nitrite cream applied per 1 cm^2 of the total ulcerated area. Areas will be rounded to the nearest 1 cm^2. If a participant has more than one ulcer, all of them will be treated with either "study cream" in this intervention.
Period: Overall Study
Arm/Group | Placebo | Topical Sodium Nitrite
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: For this study, the fundamental analysis unit was the participant and not the ulcer(s). All data is presented accordingly.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Topical Sodium Nitrite | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.0) | 47.6 (13.8) | 43.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 7 | 17
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18
Total Ulcerated Surface Area [Mean (Standard Deviation); unit: cm^2] — Surface area measurements of the ulcer(s) were obtained and photographed with defined lighting, distance, exposure, and camera type. Total ulcerated surface area measurements were obtained using digital planimetry and measuring the longest length and widest width of the ulcer. Results are summarized by study arm using basic descriptive statistics and reported in cm^2.
  cm^2 | 11.4 (12.3) | 16.6 (15.4) | 13.7 (13.6)
Sickle Cell Genotype [Count of Participants; unit: Participants] — Sickle cell genotype confirmation was confirmed by hemoglobin electrophoresis analysis at baseline or patient charts. Participants were categorized as either:
  HbSS: Homozygous sickle cell disease, considered the most severe form; HbSB+: Hemoglobin S-beta thalassemia, a compound heterozygous condition considered a milder form; HbSC: 2nd most common variant and a milder form; HbSD: a double heterozygous state of two mutant alleles; or HbS/O(Arab): a rare compound heterozygous variant
  The number/percentage of each genotype is summarized and reported by study arm.
  Participants
    HbSS | 10 | 7 | 17
    HbSB+ | 0 | 1 | 1
    HbSC | 0 | 0 | 0
    HbSD | 0 | 0 | 0
    HbS/O (Arab) | 0 | 0 | 0
Hydroxyurea Usage [Count of Participants; unit: Participants] — The number/percentage of participants actively using Hydroxyurea (a disease-modifying agent) at baseline was evaluated. Hydroxyurea usage was confirmed and reported using a dichotomous "Yes" or "No" assessment.
  Participants
    No | 4 | 5 | 9
    Yes | 6 | 3 | 9
Methemoglobin Levels [Mean (Standard Deviation); unit: percentage of total hemoglobin] — Samples were collected and analyzed by co-oximetry to determine Methemoglobin (metHb) levels in order to exclude participants with congenital methemoglobinemia. Patients who had at least two documented metHb levels below the 3.5% threshold continued the study even if the meth Hb levels elevated above 3.5% during the weeks leading to the first application, as long as they remain below 4.5%. Baseline results are summarized by study arm using basic descriptive statistics and results were expressed as a percentage of the total hemoglobin in the sample.
  percentage of total hemoglobin | 1.76 (0.635) | 1.49 (0.698) | 1.64 (0.658)
Visual Analog Scale (VAS) for Pain Intensity [Mean (Standard Deviation); unit: score on a scale] — The Visual Analog Scale (VAS) was used to assess existing pain intensity prior to the initiation of treatment. The VAS is a pain intensity scale that uses a 10-centimeter (cm) line where 0 represents "No pain" and 10 represents "Worst possible pain." Participants were asked to mark current pain levels on the line and the distance from the "No pain" end of the line measured in cm was used to determine a VAS score. VAS scores were summarized by study arm/group using basic descriptive statistics. Higher scores were associated with greater overall pain intensity.
  score on a scale | 5.3 (2.49) | 4.28 (1.62) | 4.84 (2.15)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Tolerability (Methemoglobin Level)
Description: Assessment of tolerability was determined by evaluating the change in methemoglobin level from baseline through the end of study at week 10. Samples were collected and Methemoglobin levels were measured by co-oximetry Results are summarized by study arm using basic descriptive statistics and expressed as a percentage of the total hemoglobin in the sample.
Time Frame: Baseline through last available measurement, up to 10 weeks
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: percentage of total hemoglobin
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
percentage of total hemoglobin | -0.05 [-0.6 to 0.4] | 0.25 [-0.3 to 0.4]
Statistical Analysis 1: Comparison: Placebo vs Topical Sodium Nitrite; Change in methemoglobin from baseline to end of study (EOS) for all participants; Test type: Superiority; p = 0.2967, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in methemoglobin at baseline and EOS for all participants between treatment arms using a Wilcoxon signed rank test

2. Primary Outcome: Change in Total Ulcerated Surface Area
Description: Change in total ulcerated surface area from baseline was assessed through the last study visit at 10 weeks. Surface area measurements of the ulcer were obtained and photographed with defined lighting, distance, exposure, and camera type. Total ulcerated surface area measurements were obtained using digital planimetry and measuring the longest length and widest width of the ulcer(s). Results are summarized by study arm using basic descriptive statistics and reported in cm^2. Negative results are indicative of a reduction in group median total ulcerated surface area from baseline and positive results are indicative of an increase in group median total ulcerated surface area from baseline.
Time Frame: From Baseline through last study visit at 10 weeks
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
cm^2 | -1.50 [-3.90 to -0.068] | -3.26 [-12.0 to 0.987]
Statistical Analysis 1: Comparison: Placebo vs Topical Sodium Nitrite; Change in total ulcerated surface area from baseline to end of study (EOS); Test type: Superiority; p = 0.2818, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in total ulcerated surface area at baseline and EOS between treatment arms using a Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Placebo vs Topical Sodium Nitrite; Difference in frequency of 25% total ulcerated surface area reduction between treatment arms; Test type: Superiority; p = 1.0, Fisher Exact; Fisher's exact test was used to test for differences in frequencies between treatment arms

3. Primary Outcome: Change in Ulcer Pain
Description: Change in Ulcer Pain from baseline through the last study visit at 10 weeks were assessed using the Visual Analog Scale (VAS). The VAS is a widely used tool to quantify subjective pain perception over time and in this study was used to determine the efficacy of the topical sodium nitrite. Participants were asked to mark a point on a line indicating the severity of their pain on a 0-10 scale, with "0" representing "No pain" and "10" representing the "Worst possible pain." A decrease in VAS score is indicative of a reduction in ulcer pain. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From Baseline through last study visit at 10 weeks
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
score on a scale | -0.5 [-2.7 to 1.2] | 0.9 [-3.8 to 2.6]
Statistical Analysis 1: Comparison: Placebo vs Topical Sodium Nitrite; Change in average pain from baseline to end of study (EOS); Test type: Superiority; p = 0.3754, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in average pain at baseline and EOS between treatment arms using a Wilcoxon signed rank test

4. Primary Outcome: Number of Participants With Total Ulcerated Surface Area Reduction
Description: The number of participants who achieved an objective reduction in total surface area of the ulcer of >= 25% from baseline is summarized and reported as a dichotomous ("No" or "Yes") variable.
Time Frame: From Baseline through last study visit at 10 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
Participants
  No | 5 | 4
  Yes | 5 | 4

5. Secondary Outcome: Hydroxyurea Effect on Assessment of Tolerability
Description: Hydroxyurea effect on Assessment of Tolerability, as determined by the change in Methemoglobin level, was conducted to evaluate the effect of hydroxyurea in combination with the topical sodium nitrite or placebo. Samples were collected and Methemoglobin levels were measured by co-oximetry. Study outcomes between participants with use of ("HU") and non-use of ("No HU") hydroxyurea are summarized as an increased or decreased percentage by study arm and analyzed using Wilcoxon-Mann-Whitney statistical testing.
Time Frame: From Baseline through last study visit at 10 weeks
Population: Number of participants analyzed identified in table below. For this study, the fundamental analysis unit was the participant and not the ulcer(s). All data is presented accordingly.
Measure: Median (Inter-Quartile Range); unit: percentage of total hemoglobin
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
percentage of total hemoglobin
  HU: number analyzed (Participants) | 5 | 3
  HU | -0.6 [-0.7 to -0.4] | 0.2 [0 to 0.3]
  No HU: number analyzed (Participants) | 5 | 5
  No HU | 0.3 [0 to 0.5] | 0.3 [-0.6 to 0.5]
Statistical Analysis 1: Comparison: Placebo vs Topical Sodium Nitrite; Change in methemoglobin from baseline to end of study (EOS) for participants on Hydroxyurea (HU); Test type: Superiority; p = 0.1165, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in methemoglobin at baseline and EOS between treatment arms for participants on Hydroxyurea (HU) using a Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Placebo vs Topical Sodium Nitrite; Change in methemoglobin from baseline to end of study (EOS) for participants off Hydroxyurea (HU); Test type: Superiority; p = 0.4583, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in methemoglobin at baseline and EOS between treatment arms for participants off Hydroxyurea (HU) using a Wilcoxon signed rank test

6. Secondary Outcome: Hydroxyurea Effect on Change in Total Ulcerated Surface Area
Description: Hydroxyurea effect on Change in Total Ulcerated Surface Area was conducted to evaluate the effect of hydroxyurea in combination with the topical sodium nitrite or placebo. Surface area measurements of the ulcer were obtained and photographed with defined lighting, distance, exposure, and camera type. Total ulcerated surface area measurements were obtained using digital planimetry and measuring the longest length and widest width of the ulcer(s). Study outcomes between participants with use of ("HU") and non-use of ("No HU") hydroxyurea are summarized by study arm as an increase or decrease in total ulcerated surface area in cm^2 and analyzed using Wilcoxon-Mann-Whitney and Fisher Exact statistical testing. Negative results are indicative of a reduction in group median total ulcerated surface area from baseline and positive results are indicative of an increase in group median total ulcerated surface area from baseline (with or without Hydroxyurea).
Time Frame: From Baseline through last study visit at 10 weeks
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
cm^2
  HU: number analyzed (Participants) | 5 | 3
  HU | -1.34 [-1.592 to -0.068] | -3.506 [-6.97 to -3.013]
  No HU: number analyzed (Participants) | 5 | 5
  No HU | -2.081 [-3.897 to -1.412] | -0.57 [-17.04 to 2.031]
Statistical Analysis 1: Comparison: Placebo vs Topical Sodium Nitrite; Change in total ulcerated surface area from baseline to end of study (EOS) for participants on Hydroxyurea (HU); Test type: Superiority; p = 0.068, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in total ulcerated surface area at baseline and EOS between treatment arms for participants on Hydroxyurea (HU) using a Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Placebo vs Topical Sodium Nitrite; Change in total ulcerated surface area from baseline to end of study (EOS) for participants off Hydroxyurea (HU); Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in total ulcerated surface area at baseline and EOS between treatment arms for participants off Hydroxyurea (HU) using a Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Placebo vs Topical Sodium Nitrite; Difference in frequency of 25% total ulcerated surface area reduction between treatment arms for participants on Hydroxyurea (HU); Test type: Superiority; p = 1.0, Fisher Exact; Difference in frequency of 25% total ulcerated surface area reduction between treatment arms for participants on Hydroxyurea (HU)
Statistical Analysis 4: Comparison: Placebo vs Topical Sodium Nitrite; Difference in frequency of 25% total ulcerated surface area reduction between treatment arms for participants off Hydroxyurea (HU); Test type: Superiority; p = 1.0, Fisher Exact; Fisher's exact test was used to test for differences in frequencies between treatment arms for participants off Hydroxyurea (HU)

7. Secondary Outcome: Hydroxyurea Effect on Change in Ulcer Pain
Description: Hydroxyurea effect on change in Ulcer Pain was conducted to evaluate the effect of hydroxyurea in combination with the topical sodium nitrite or placebo. Ulcer pain assessments were conducted using the Visual Analog Scale (VAS). The VAS is used to quantify subjective pain perception over time and in this study was used to determine the efficacy of the topical sodium nitrite. Participants were asked to mark a point on a line indicating the severity of their pain on a 0-10 scale, with "0" representing "No pain" and "10" representing the "Worst possible pain." Study outcomes between participants with use of ("HU") and non-use of ("No HU") hydroxyurea are summarized by study arm as an increase or decrease in ulcer pain and analyzed using Wilcoxon-Mann-Whitney statistical testing. Negative results are indicative of a decrease in group median ulcer pain from baseline and positive results are indicative of an increase in group median ulcer pain from baseline (with or without Hydroxyurea).
Time Frame: From Baseline through last study visit at 10 weeks
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Topical Sodium Nitrite
Number analyzed (Participants) | 10 | 8
score on a scale
  HU: number analyzed (Participants) | 5 | 3
  HU | 0.35 [-1.25 to 2.10] | 0.9 [-5.0 to 2.4]
  No HU: number analyzed (Participants) | 5 | 5
  No HU | -2.70 [-4.0 to 0.0] | 1.0 [-2.2 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs Topical Sodium Nitrite; Change in average pain from baseline to end of study (EOS) for participants on Hydroxyurea (HU); Test type: Superiority; p = 0.4298, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in average pain at baseline and EOS between treatment arms for participants on Hydroxyurea (HU) using a Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Placebo vs Topical Sodium Nitrite; Change in average pain from baseline to end of study (EOS) for participants off Hydroxyurea (HU); Test type: Superiority; p = 0.2701, Wilcoxon (Mann-Whitney) — A matched pairs design was employed to test for changes in average pain at baseline and EOS between treatment arms for participants off Hydroxyurea (HU) using a Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Arm/Group | Placebo | Topical Sodium Nitrite
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/8
Other Adverse Events (participants affected / at risk) | 9/10 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Topical Sodium Nitrite (N=8)
Vaso-occlusive Crisis (General disorders) | 3 (4) | 2 (7) — Sickle cell pain/Vaso-occlusive pain noted in all Topical Sodium Nitrite patients and 2 of 3 Placebo patients (other patient documented with nonspecific Pain, hospitalization indicated).
Ulcer Infection (Infections and infestations) | 0 (0) | 1 (1) — Verbatim Term: Wound Infection. Hospitalization indicated
Acute Myeloid Leukemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Topical Sodium Nitrite (N=8)
Vaso-occlusive Crisis (General disorders) | 0 | 3 — Verbatim Terms: Sickle cell pain/Vaso-occlusive crisis/Ulcer Pain
Headache (Nervous system disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Left-sided
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Ulcer Infection (Infections and infestations) | 2 | 1 — Verbatim Terms: Wound Infection or Ulcer Infection
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Abnormal Blood Smear (Blood and lymphatic system disorders) | 1 | 0 — Laboratory result indicating blast on Complete Blood Count (CBC) report
Critical Low Lab Value (Investigations) | 1 | 0 — Verbatim Term cited
Palpitations (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Body Ache (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, enrollment in the clinical trial did not reach the target number of participants needed to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT02863068/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT02863068/ICF_001.pdf